CLINICAL TRIAL: NCT03232307
Title: A Phase II Study of Ibrutinib Plus Rituximab and Lenalidomide in Elderly Patients With Newly Diagnosed MCL
Brief Title: Ibrutinib Plus Rituximab and Lenalidomide in Treating Elderly Participants With Newly Diagnosed Mantle Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor does not wish to proceed
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0280; NCI-2018-01271 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0280 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: CCND1 Positive; CD20-Positive Neoplastic Cells Present; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ibrutinib; Lenalidomide; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, rituximab, lenalidomide, dexamethasone) (Experimental): Participants receive ibrutinib PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Participants also receive rituximab IV on days 1, 8, 15 and 22 in course 1 and 2, on day 1 of course 3-8, and then on day 1 of every other 28-day course, lenalidomide PO on days 1-21, and dexamethasone PO weekly. Treatment with rituximab repeats every 28 days for 2 years, with lenalidomide for 1 year, and with dexamethasone for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Ibrutinib; Drug: Lenalidomide; Biological: Rituximab

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83

SUMMARY:
This phase II trial studies how well ibrutinib plus rituximab and lenalidomide work in treating elderly participants with newly diagnosed mantle cell lymphoma. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as rituximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ibrutinib plus rituximab and lenalidomide may work better in treating elderly participants with newly diagnosed mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall response rate (ORR) at 4 months of ibrutinib plus rituximab and lenalidomide in elderly patients with newly-diagnosed, untreated mantle cell lymphoma (MCL).

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile of the combination of ibrutinib plus rituximab and lenalidomide in newly diagnosed, untreated MCL.

II. To estimate the overall response rate (ORR); (partial response [PR] or better), the response duration (DOR), progression-free survival (PFS), time to progression (TTP) and overall survival (OS). Clinical benefit response [(CBR) = marginal response (MR) + ORR] will also be evaluated.

EXPLORATORY OBJECTIVES:

I. Correlative studies will be aimed at confirming the mechanism of action of the combination and to identify predictors of response or resistance to therapy.

OUTLINE:

Participants receive ibrutinib orally (PO) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Participants also receive rituximab intravenously (IV) on days 1, 8, 15 and 22 in course 1 and 2, on day 1 of course 3-8, and then on day 1 of every other 28-day course, lenalidomide PO on days 1-21, and dexamethasone PO weekly. Treatment with rituximab repeats every 28 days for 2 years, with lenalidomide for 1 year, and with dexamethasone for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days, every 3 months for 1 year, and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MCL with CD20 and cyclin D1 positivity in tissue biopsy.
* Ki-67 >= 50%.
* Patients must have never received any prior systemic therapy for their disease.
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Patients should in general have bi-dimensional measurable disease using the Cheson criteria (measurable disease by computed tomography [CT] scan defined as at least 1 lesion that measures >= 1.5 cm in single dimension) (bone marrow or gastrointestinal [GI] only involvement is acceptable).
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less.
* Absolute neutrophil count (ANC) >= 1000/mm^3 without transfusion support.
* Platelet count > 100,000/mm^3. Patients who have bone marrow infiltration by MCL are eligible if their platelet level is >= 50,000 /mm^3 independent of platelet transfusions.
* Aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) =< 3 x upper limit of normal.
* Serum bilirubin < 1.5 mg/dl unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin.
* Creatinine (Cr) clearance >= 25 mL/min (per Cockcroft-Gault equation).
* Disease free of prior malignancies of equal to or greater than 6 months with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or other malignancies in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated, with a life expectancy > 3 years.
* Patients must be willing to receive transfusions of blood products.
* Willing and able to participate in all study related procedures and therapy including swallowing capsules without difficulty.
* Men must agree 1) to use a latex condom during sexual contact with a female of childbearing potential (FCBP) even if they have had a vasectomy from the time of signing the informed consent form through 90 days after the last dose of lenalidomide and ibrutinib; 2) to not donate sperm during and after the study. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide through 90 days and ibrutinib through 30 days after the last dose of study drug. FCBP must also agree to ongoing pregnancy testing.
* All patients must be registered in and must comply with all requirements of the Revlimid Rems program.

Exclusion Criteria:

* Any serious medical condition that, in the investigator opinion, places the patient at unacceptable risk and/or would prevent the subject from signing the informed consent form. Examples include but are not limited to, uncontrolled hypertension, uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, active infection requiring treatment with intravenous (IV) antibiotics, antiviral or antifungal agents, active hemorrhage, or psychiatric illness in the investigator's opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form.
* Pregnant or breastfeeding females.
* Known human immunodeficiency virus (HIV) infection. Patients with active hepatitis B infection (not including patients with prior hepatitis B vaccination; or positive serum hepatitis B antibody). Known hepatitis C infection is allowed as long as there is no active disease. These patients should be optimized by GI consultation for hepatitis B and infectious disease consult for hepatitis C.
* The patient has a prior or concurrent malignancy that in the opinion of the investigator, presents a greater risk to the patient's health and survival, than of the MCL, within the subsequent 6 months at the time of consent.
* History of stroke or intracranial hemorrhage within 6 months prior to signing the consent.
* Patients at high-risk for thromboembolic disease, such as those with prior heterotopic ossification (h/o) deep venous thrombosis (DVT).
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within 6 months at the time of consent or any class 3 (moderate) or 4 (severe) cardiac disease defined by the New York Heart Association classification.
* Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular block (AV block) type II, 3rd degree block, bradycardia (< 50 beats per minute [bpm]), or corrected QT (QTc) > 500 msec.
* Patients with persistent and uncontrolled atrial fibrillation even if rate controlled.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Major surgery or wound that has not fully healed within 4 weeks or vaccination with live attenuated vaccines within 4 weeks of the first dose of study drugs.
* Requires concomitant anticoagulation with warfarin or equivalent vitamin K antagonist.
* Requires treatment with strong cytochrome P4503A (CYP3A) inhibitors.
* All patients with central nervous system lymphoma.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) per International Workshop Standardization Response Criteria for non-Hodgkin's lymphoma | At 4 months (each cycle is 28 days)
  The overall response (complete response + partial response) at four months and toxicity at one month (during course 1) will be monitored simultaneously using the Bayesian approach of Thall, Simon, Estey as extended by Thall and Sung. Independence was assumed between or and toxicity, where toxicity is defined as dose-limiting toxicity (DLT) within cycle 1.

SECONDARY OUTCOMES:
Incidence of adverse events per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.03 | At 1 month (cycle 1 is 28 days)
  Toxicity data by type and severity will be summarized by frequency tables. For the efficacy endpoints, intend-to-treat analysis will be performed. For the toxicity endpoint, per-treated analysis will be performed to include any patient who received the treatment regardless of the eligibility nor the duration or dose of the treatment received.
Overall survival (OS) | Up to 4 years
  Summary statistics will be provided for continuous variables. Frequency tables will be used to summarize categorical variables. The distribution of time-to-event endpoints including overall survival and progression free survival will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Cox proportional hazard regression will be employed for multivariate analysis on time-to-event outcomes.
Progression-free survival | Up to 4 years
  Summary statistics will be provided for continuous variables. Frequency tables will be used to summarize categorical variables. The distribution of time-to-event endpoints including overall survival and progression free survival will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Cox proportional hazard regression will be employed for multivariate analysis on time-to-event outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org